CLINICAL TRIAL: NCT01872962
Title: Prospective Randomized Trial Comparing Concurrent Chemoradiotherapy With or Without Induction Gemcitabine and Cisplatin in Patients With Locoregionally Advanced Nasopharyngeal Carcinoma
Brief Title: Induction Gemcitabine and Cisplatin in Patients With Locoregionally Advanced Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Fudan University (Other); West China Hospital (Other); Tongji Hospital (Other); Peking University (Other); Zhejiang Cancer Hospital (Other); First People's Hospital of Foshan (Other); Cancer Hospital of Guangxi Medical University (Other); Jiangxi Provincial Cancer Hospital (Other); Xijing hospital of The fourth military medical university (Unknown); Cancer Hospital of Guizhou Province (Other); Affiliated Cancer Hospital of Shantou University Medical College (Other); Fifth Affiliated Hospital, Sun Yat-Sen University (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Jun Ma, MD, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2013-022-01
Record Dates: First submitted 2013-05-31; First posted 2013-06-07 (Estimated); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal carcinoma; Induction chemotherapy; Concurrent chemoradiotherapy; Clinical trial
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Gemcitabine; Cisplatin; Induction Chemotherapy; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Induction chemotherapy+IMRT and concurrent cisplatin (Experimental): Patients receive gemcitabine (1000 mg/m² d1,8) and cisplatin (80mg/m² d1) every 3 weeks for 3 cycles before radiotherapy, and then receive intensity modulated-radiotherapy (IMRT), concurrently with cisplatin 100 mg/m² every 3 weeks for 3 cycles.
  Interventions: Drug: gemcitabine and cisplatin (Induction chemotherapy); Radiation: IMRT and concurrent cisplatin
- IMRT and concurrent cisplatin (Active Comparator): Patients receive intensity modulated-radiotherapy (IMRT), concurrently with cisplatin 100 mg/m² every 3 weeks for 3 cycles.
  Interventions: Radiation: IMRT and concurrent cisplatin

INTERVENTIONS:
Drug: gemcitabine and cisplatin (Induction chemotherapy) — Patients receive gemcitabine (1000 mg/m² d1,8) and cisplatin (80mg/m² d1) every 3 weeks for 3 cycles before concurrent chemoradiotherapy.
  Other Names: gemcitabine and cisplatin (GP)
  Arms: Induction chemotherapy+IMRT and concurrent cisplatin
Radiation: IMRT and concurrent cisplatin — Intensity modulated-radiotherapy (IMRT) is given as 2.0-2.30 Gy per fraction with five daily fractions per week for 6-7 weeks to a total dose of 66 Gy or greater to the primary tumor, concurrently with cisplatin 100 mg/m² every 3 weeks for 3 cycles.

SUMMARY:
The purpose of this study is to compare induction chemotherapy (gemcitabine+cisplatin) plus concurrent chemoradiotherapy (CCRT) with CCRT alone in patients with locoregionally advanced nasopharyngeal carcinoma(NPC), in order to confirm the value of induction chemotherapy in NPC patients.

DETAILED DESCRIPTION:
Patients Patients with non-keratinizing NPC T3-4N1M0/TxN2-3M0 (UICC/AJCC 7th edition) are randomly assigned to receive induction chemotherapy plus CCRT or CCRT alone. Patients in both groups receive cisplatin 100 mg/m² every 3 weeks for 3 cycles, concurrently with intensity-modulated radiotherapy (IMRT). IMRT is given as 2.0-2.30 Gy per fraction with five daily fractions per week for 6-7 weeks to a total dose of 66 Gy or greater to the primary tumor. The induction chemotherapy plus CCRT group receive gemcitabine (1000 mg/m² d1,8) and cisplatin (80mg/m² d1) every 3 weeks for three cycles before CCRT. Our primary endpoint is failure-free survival(FFS). Secondary end points include overall survival (OS), locoregional failure-free survival (LR-FFS), distant failure-free survival (D-FFS) rates and toxic effects. All efficacy analyses are conducted in the intention-to-treat population, and the safety population include only patients who receive their randomly assigned treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly histologically confirmed non-keratinizing (according to WHO histologically type).
* Tumor staged as T3-4N1/N2-3 (according to the 7th AJCC edition).
* No evidence of distant metastasis (M0).
* Satisfactory performance status: Karnofsky scale (KPS) ≥ 70.
* Adequate marrow: leucocyte count ≥ 4000/μL, hemoglobin ≥ 90g/L and platelet count ≥ 100000/μL.
* Normal liver function test: Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST) < 1.5×upper limit of normal (ULN) concomitant with alkaline phosphatase (ALP) ≤ 2.5×ULN, and bilirubin ≤ ULN.
* Adequate renal function: creatinine clearance ≥ 60 ml/min.
* Patients must be informed of the investigational nature of this study and give written informed consent.

Exclusion Criteria:

* WHO Type keratinizing squamous cell carcinoma or basaloid squamous cell carcinoma.
* Age > 65 or < 18.
* Treatment with palliative intent.
* Prior malignancy except adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer.
* Pregnancy or lactation (consider pregnancy test in women of child-bearing age and emphasize effective contraception during the treatment period).
* History of previous RT (except for non-melanomatous skin cancers outside intended RT treatment volume).
* Prior chemotherapy or surgery (except diagnostic) to primary tumor or nodes.
* Any severe intercurrent disease, which may bring unacceptable risk or affect the compliance of the trial, for example, unstable cardiac disease requiring treatment, renal disease, chronic hepatitis, diabetes with poor control (fasting plasma glucose > 1.5×ULN), and emotional disturbance.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 2013-11; Primary Completion 2018-11 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Failure-free survival | 3-year
  Failure-free survival rate is calculated from the date of randomization to the date of treatment failure or death from any cause, whichever is first.

SECONDARY OUTCOMES:
Overall survival | 3-year
  Overall survival is calculated from randomization to death from any cause.
Locoregional failure-free survival | 3-year
  Locoregional failure-free survival is calculated from randomization to the first locoregional failure.
Distant failure-free survival | 3-year
  Distant failure-free survival is calculated from randomization to the first remote failure.
Number of participants with adverse events | up to 3 years
  Incidence of acute and late toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Jun Ma, M.D., Study Chair — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Jemal A, Bray F, Center MM, Ferlay J, Ward E, Forman D. Global cancer statistics. CA Cancer J Clin. 2011 Mar-Apr;61(2):69-90. doi: 10.3322/caac.20107. Epub 2011 Feb 4. PMID 21296855
- [Background] Edge SB, Byrd DR, Compton CC, et al: AJCC Cancer Staging Manual (ed 7th). New York, Springer, 2010
- [Background] Lai SZ, Li WF, Chen L, Luo W, Chen YY, Liu LZ, Sun Y, Lin AH, Liu MZ, Ma J. How does intensity-modulated radiotherapy versus conventional two-dimensional radiotherapy influence the treatment results in nasopharyngeal carcinoma patients? Int J Radiat Oncol Biol Phys. 2011 Jul 1;80(3):661-8. doi: 10.1016/j.ijrobp.2010.03.024. Epub 2010 Jul 17. PMID 20643517
- [Background] Baujat B, Audry H, Bourhis J, Chan AT, Onat H, Chua DT, Kwong DL, Al-Sarraf M, Chi KH, Hareyama M, Leung SF, Thephamongkhol K, Pignon JP; MAC-NPC Collaborative Group. Chemotherapy in locally advanced nasopharyngeal carcinoma: an individual patient data meta-analysis of eight randomized trials and 1753 patients. Int J Radiat Oncol Biol Phys. 2006 Jan 1;64(1):47-56. doi: 10.1016/j.ijrobp.2005.06.037. PMID 16377415
- [Background] Langendijk JA, Leemans CR, Buter J, Berkhof J, Slotman BJ. The additional value of chemotherapy to radiotherapy in locally advanced nasopharyngeal carcinoma: a meta-analysis of the published literature. J Clin Oncol. 2004 Nov 15;22(22):4604-12. doi: 10.1200/JCO.2004.10.074. PMID 15542811
- [Background] International Nasopharynx Cancer Study Group; VUMCA I Trial. Preliminary results of a randomized trial comparing neoadjuvant chemotherapy (cisplatin, epirubicin, bleomycin) plus radiotherapy vs. radiotherapy alone in stage IV(> or = N2, M0) undifferentiated nasopharyngeal carcinoma: a positive effect on progression-free survival. Int J Radiat Oncol Biol Phys. 1996 Jun 1;35(3):463-9. doi: 10.1016/s0360-3016(96)80007-1. PMID 8655368
- [Background] Chua DT, Sham JS, Choy D, Lorvidhaya V, Sumitsawan Y, Thongprasert S, Vootiprux V, Cheirsilpa A, Azhar T, Reksodiputro AH. Preliminary report of the Asian-Oceanian Clinical Oncology Association randomized trial comparing cisplatin and epirubicin followed by radiotherapy versus radiotherapy alone in the treatment of patients with locoregionally advanced nasopharyngeal carcinoma. Asian-Oceanian Clinical Oncology Association Nasopharynx Cancer Study Group. Cancer. 1998 Dec 1;83(11):2270-83. PMID 9840526
- [Background] Ma J, Mai HQ, Hong MH, Min HQ, Mao ZD, Cui NJ, Lu TX, Mo HY. Results of a prospective randomized trial comparing neoadjuvant chemotherapy plus radiotherapy with radiotherapy alone in patients with locoregionally advanced nasopharyngeal carcinoma. J Clin Oncol. 2001 Mar 1;19(5):1350-7. doi: 10.1200/JCO.2001.19.5.1350. PMID 11230478
- [Background] Hareyama M, Sakata K, Shirato H, Nishioka T, Nishio M, Suzuki K, Saitoh A, Oouchi A, Fukuda S, Himi T. A prospective, randomized trial comparing neoadjuvant chemotherapy with radiotherapy alone in patients with advanced nasopharyngeal carcinoma. Cancer. 2002 Apr 15;94(8):2217-23. doi: 10.1002/cncr.10473. PMID 12001120
- [Background] Barton-Burke M. Gemcitabine: a pharmacologic and clinical overview. Cancer Nurs. 1999 Apr;22(2):176-83. doi: 10.1097/00002820-199904000-00011. PMID 10217035
- [Background] Foo KF, Tan EH, Leong SS, Wee JT, Tan T, Fong KW, Koh L, Tai BC, Lian LG, Machin D. Gemcitabine in metastatic nasopharyngeal carcinoma of the undifferentiated type. Ann Oncol. 2002 Jan;13(1):150-6. doi: 10.1093/annonc/mdf002. PMID 11865813
- [Background] Ma BB, Tannock IF, Pond GR, Edmonds MR, Siu LL. Chemotherapy with gemcitabine-containing regimens for locally recurrent or metastatic nasopharyngeal carcinoma. Cancer. 2002 Dec 15;95(12):2516-23. doi: 10.1002/cncr.10995. PMID 12467065
- [Background] Zhang L, Zhang Y, Huang PY, Xu F, Peng PJ, Guan ZZ. Phase II clinical study of gemcitabine in the treatment of patients with advanced nasopharyngeal carcinoma after the failure of platinum-based chemotherapy. Cancer Chemother Pharmacol. 2008 Jan;61(1):33-8. doi: 10.1007/s00280-007-0441-8. Epub 2007 Mar 20. PMID 17909810
- [Background] Ngan RK, Yiu HH, Lau WH, Yau S, Cheung FY, Chan TM, Kwok CH, Chiu CY, Au SK, Foo W, Law CK, Tse KC. Combination gemcitabine and cisplatin chemotherapy for metastatic or recurrent nasopharyngeal carcinoma: report of a phase II study. Ann Oncol. 2002 Aug;13(8):1252-8. doi: 10.1093/annonc/mdf200. PMID 12181249
- [Background] Jiang Y, Wei YQ, Luo F, Zou LQ, Liu JY, Peng F, Huang MJ, He QM. Gemcitabine and cisplatin in advanced nasopharyngeal carcinoma: a pilot study. Cancer Invest. 2005;23(2):123-8. PMID 15813504
- [Background] Yau TK, Lee AW, Wong DH, Yeung RM, Chan EW, Ng WT, Tong M, Soong IS. Induction chemotherapy with cisplatin and gemcitabine followed by accelerated radiotherapy and concurrent cisplatin in patients with stage IV(A-B) nasopharyngeal carcinoma. Head Neck. 2006 Oct;28(10):880-7. doi: 10.1002/hed.20421. PMID 16721741
- [Background] He X, Ou D, Ying H, Zhu G, Hu C, Liu T. Experience with combination of cisplatin plus gemcitabine chemotherapy and intensity-modulated radiotherapy for locoregionally advanced nasopharyngeal carcinoma. Eur Arch Otorhinolaryngol. 2012 Mar;269(3):1027-33. doi: 10.1007/s00405-011-1669-9. Epub 2011 Jun 26. Erratum In: Eur Arch Otorhinolaryngol. 2012 Mar;269(3):1035. Xiayun, He [corrected to He, Xiayun]. PMID 21706324
- [Background] Freedman J, Furberg C, DeMets D: Fundamentals of clinical trials. New York, Springer-Verlag, 1998
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Cox JD, Stetz J, Pajak TF. Toxicity criteria of the Radiation Therapy Oncology Group (RTOG) and the European Organization for Research and Treatment of Cancer (EORTC). Int J Radiat Oncol Biol Phys. 1995 Mar 30;31(5):1341-6. doi: 10.1016/0360-3016(95)00060-C. No abstract available. PMID 7713792
- [Background] Chow SC, Shao J, Wang H: Sample Size Calculations in Clinical Research. New York, Marcel Dekker, 2003
- [Derived] Lv J, Wei Y, Yin JH, Chen YP, Zhou GQ, Wei C, Liang XY, Zhang Y, Zhang CJ, He SW, He QM, Huang ZL, Guan JL, Shen JY, Li XM, Li JY, Li WF, Tang LL, Mao YP, Guo R, Sun R, Zheng YH, Zhou WW, Xiong KX, Wang SQ, Jin X, Liu N, Li GB, Kuang DM, Sun Y, Ma J. The tumor immune microenvironment of nasopharyngeal carcinoma after gemcitabine plus cisplatin treatment. Nat Med. 2023 Jun;29(6):1424-1436. doi: 10.1038/s41591-023-02369-6. Epub 2023 Jun 6. PMID 37280275
- [Derived] Zhang Y, Chen L, Hu GQ, Zhang N, Zhu XD, Yang KY, Jin F, Shi M, Chen YP, Hu WH, Cheng ZB, Wang SY, Tian Y, Wang XC, Sun Y, Li JG, Li WF, Li YH, Mao YP, Zhou GQ, Sun R, Liu X, Guo R, Long GX, Liang SQ, Li L, Huang J, Long JH, Zang J, Liu QD, Zou L, Su QF, Zheng BM, Xiao Y, Guo Y, Han F, Mo HY, Lv JW, Du XJ, Xu C, Liu N, Li YQ, Xie FY, Sun Y, Ma J, Tang LL. Final Overall Survival Analysis of Gemcitabine and Cisplatin Induction Chemotherapy in Nasopharyngeal Carcinoma: A Multicenter, Randomized Phase III Trial. J Clin Oncol. 2022 Aug 1;40(22):2420-2425. doi: 10.1200/JCO.22.00327. Epub 2022 Jun 16. PMID 35709465
- [Derived] Xu C, Yang KB, Feng RJ, Chen L, Du XJ, Mao YP, Li WF, Liu Q, Sun Y, Ma J. Radiotherapy interruption due to holidays adversely affects the survival of patients with nasopharyngeal carcinoma: a joint analysis based on large-scale retrospective data and clinical trials. Radiat Oncol. 2022 Feb 19;17(1):36. doi: 10.1186/s13014-022-02006-5. PMID 35183221
- [Derived] Zhang Y, Chen L, Hu GQ, Zhang N, Zhu XD, Yang KY, Jin F, Shi M, Chen YP, Hu WH, Cheng ZB, Wang SY, Tian Y, Wang XC, Sun Y, Li JG, Li WF, Li YH, Tang LL, Mao YP, Zhou GQ, Sun R, Liu X, Guo R, Long GX, Liang SQ, Li L, Huang J, Long JH, Zang J, Liu QD, Zou L, Su QF, Zheng BM, Xiao Y, Guo Y, Han F, Mo HY, Lv JW, Du XJ, Xu C, Liu N, Li YQ, Chua MLK, Xie FY, Sun Y, Ma J. Gemcitabine and Cisplatin Induction Chemotherapy in Nasopharyngeal Carcinoma. N Engl J Med. 2019 Sep 19;381(12):1124-1135. doi: 10.1056/NEJMoa1905287. Epub 2019 May 31. PMID 31150573
- [Derived] Chua ML, Chan AT. Gemcitabine: a game changer in nasopharyngeal carcinoma. Lancet. 2016 Oct 15;388(10054):1853-1854. doi: 10.1016/S0140-6736(16)31394-0. Epub 2016 Aug 23. No abstract available. PMID 27567280